CLINICAL TRIAL: NCT07161674
Title: WhatsApp Intervention for Seniors' Digital and Cognitive Management (WISDOM): a Mixed-methods Pilot Study
Brief Title: WhatsApp Intervention for Seniors' Digital and Cognitive Management (WISDOM)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Seah Betsy, Research Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NUS-IRB-2024-1036
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Cognition; Aged; Digital Health Literacy
Keywords: Digital health literacy; Cognitive health; Cognitive function; Older adults; Aging population; Community-based intervention; Health information seeking; Singapore; Feasibility study; Mixed methods study; WhatsApp intervention

STUDY DESIGN:
Intervention Model Description: This study uses a pilot cluster randomization design, with four active ageing centres randomized into two intervention and two control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WISDOM Intervention (Experimental): Participants in this arm will take part in the WISDOM program (WhatsApp Intervention for Seniors' Digital and cOgnitive Management). The program lasts 6 weeks and includes weekly face-to-face training sessions combined with WhatsApp-based learning activities focused on digital health literacy skills. Additional support may be offered to participants who require extra assistance.
  Interventions: Behavioral: Digital health literacy program
- Control (Usual Care) (No Intervention): Participants in this arm will continue with the usual activities provided at their active ageing centres. They will not receive the structured WISDOM program during the study period.

INTERVENTIONS:
Behavioral: Digital health literacy program — A 6-week digital health literacy program delivered through weekly face-to-face training sessions and WhatsApp activities. Additional support may be provided if needed.
  Arms: WISDOM Intervention

SUMMARY:
The goal of this clinical trial is to learn if a digital health literacy program using mobile phone chat-based application called WISDOM (WhatsApp Intervention for Seniors' Digital and cOgnitive Management) can help older adults in Singapore with fewer resources improve their digital health skills and support brain health.

The main questions it aims to answer are:

* Is it feasible to run WISDOM in senior centres, and will participants join and stay in the program?
* Does WISDOM help older adults find and use online health information?
* Does WISDOM help older adults make health decisions and impact brain functions?
* What do participants think about WISDOM, and how can it be improved?

Researchers will compare two groups:

* WISDOM group: Participants will join a 6-week program with face-to-face learning sessions and WhatsApp activities about digital health skills. Extra support will be given if needed.
* Control group: Participants will continue with their usual activities at the senior centres.

Participants in the WISDOM group will:

* Join weekly face-to-face sessions for 6 weeks
* Use WhatsApp to complete learning activities

DETAILED DESCRIPTION:
Promoting lifelong learning and digital usage are forms of cognitive stimulation that foster cognitive flexibility and connectivity with information and social networks. Functional imaging research has shown that older adults who were previously internet naïve demonstrated increased brain neural activity after learning to search online. Other studies reported that older adults who underwent in-person digital literacy programs involving internet searches, messaging, photography, and mobile application use showed improvements in overall cognition, episodic memory, and processing speed. Knowledge and skills gained through learning also promoted empowerment, psychosocial well-being, and improved quality of life.

In Singapore, formal and non-formal learning among older adults remains low, with only 13.2% participating, and those who do often have higher socioeconomic status. Socially disadvantaged older adults rarely take part, even though learning engagement has been found to improve subjective well-being more strongly in this group. Volunteer-led, one-to-one digital literacy programs for older adults with low socioeconomic status have shown promise but were resource-intensive. Thus, innovative, accessible, and affordable approaches are needed.

Chat-based applications offer a potential platform for informal learning among older adults, as they support multimedia attachments, real-time messaging, and videoconferencing. WhatsApp is a common chat-based application widely used by older adults in Singapore. Previous studies have reported positive health and behavioral outcomes of chat-based interventions in areas such as smoking cessation, diabetes, breastfeeding, and depression. However, evidence for digital health literacy interventions using mobile-based chat-based platform to promote digital health literacy skills among older adults.

This study will pilot WISDOM (WhatsApp Intervention for Seniors' Digital and cOgnitive Management) to assess feasibility and explore its potential benefits among socially disadvantaged older adults. A mixed methods design will be adopted. Four active ageing centres will be randomized into two WISDOM and two control groups. About 140 older adults with low socioeconomic status will be recruited.

The WISDOM program will last 6 weeks and include face-to-face sessions and WhatsApp-based learning. Weekly topics include, but not limited, to basics of operating search engines, websites, and mobile applications, searching online health information using Google and YouTube, evaluating the reliability of health information and applying online health information.

Participants in the WISDOM group may receive additional support where needed. A subset of participants will join qualitative interviews to share their experiences and provide feedback.

Data will be collected at three timepoints: baseline (pre-test), post-test 1 (week 7), and post-test 2 (3 months after completion) to monitor changes in digital health literacy and cognitive outcomes. Quantitative analyses will include repeated measures approaches, and qualitative data will be analyzed thematically.

This pilot study will provide insights into feasibility, acceptability, and preliminary effectiveness of WISDOM as a potentially scalable, low-resource intervention to improve digital health literacy and cognition among socially disadvantaged older adults in the community.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and above
* Own a smartphone
* Received up to primary school education or lesser
* Able to converse and read English or Mandarin

Exclusion Criteria:

* Diagnosed with dementia or at risk of dementia (MoCA) ≤ 23/24

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Digital health literacy competency | Baseline, week 7 (post-test 1), and 3 months after intervention (post-test 2).
  Competency in digital health literacy will be measured using the 21-item Digital Health Literacy Instrument (DHLI). The DHLI includes seven domains: operational skills, navigation skills, information searching, evaluating reliability, determining relevance, adding self-generated content, and protecting privacy. Internal consistency for the tool is α=0.87. In addition to the self-reported items, seven performance-based items will also be included for objective evaluation.

SECONDARY OUTCOMES:
Perceived usefulness of online health information | Baseline, week 7 (post-test 1), and 3 months after intervention (post-test 2).
  Measured using a 4-item adapted subscale from the Technology Acceptance Model 3 tool (α=0.92).
Perceived ease of using online health information | Baseline, week 7 (post-test 1), and 3 months after intervention (post-test 2).
  Measured using a 4-item adapted subscale from the Technology Acceptance Model 3 tool (α=0.93).
Attitudes towards online health information | Baseline, week 7 (post-test 1), and 3 months after intervention (post-test 2).
  Measured using a 5-item subscale of the Health Impact Questionnaire (α=0.77).
Use of online health information | Baseline, week 7 (post-test 1), and 3 months after intervention (post-test 2).
  Measured using a 4-item validated scale (α=0.82).
Changes in health behaviour and decision-making using internet-based health information | Baseline, week 7 (post-test 1), and 3 months after intervention (post-test 2).
  Measured using a modified 9-item scale assessing health behaviour change related to online health information.
Cognitive function | Baseline, week 7 (post-test 1), and 3 months after intervention (post-test 2).
  Measured using the Montreal Cognitive Assessment (MoCA), a 30-point validated screening tool for global cognition.
Cognitive domains (working memory, executive function, visuospatial coordination, psychomotor speed, attention) | Baseline, week 7 (post-test 1), and 3 months after intervention (post-test 2).
  Measured using Thinc-it, a validated computerized battery of cognitive tests. Thinc-it is not used for screening or diagnostic purposes but to explore cognition in detail.
Social support networks | Baseline, week 7 (post-test 1), and 3 months after intervention (post-test 2).
  Measured using the 6-item Abbreviated Lubben Social Network Scale, which assesses family and friend support (α=0.83).

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Seah, PhD, BSc (Nursing)(Hons), RN, Principal Investigator — National University of Singapore, Alice Lee Centre for Nursing Studies
Locations (1):
- NTUC Health Active Ageing Centre (West Cluster), Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a small pilot feasibility study involving socially disadvantaged older adults in Singapore. Sharing of IPD is not planned due to privacy, ethical, and institutional data protection requirements under Singapore's Personal Data Protection Act (PDPA). Only aggregate results will be reported in publications and presentations.

REFERENCES:
- [Background] Wang MP, Luk TT, Wu Y, Li WH, Cheung DY, Kwong AC, Lai V, Chan SS, Lam TH. Chat-based instant messaging support integrated with brief interventions for smoking cessation: a community-based, pragmatic, cluster-randomised controlled trial. Lancet Digit Health. 2019 Aug;1(4):e183-e192. doi: 10.1016/S2589-7500(19)30082-2. Epub 2019 Jul 31. PMID 33323188
- [Background] Tian Y, Zhang S, Huang F, Ma L. Comparing the Efficacies of Telemedicine and Standard Prenatal Care on Blood Glucose Control in Women With Gestational Diabetes Mellitus: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 May 25;9(5):e22881. doi: 10.2196/22881. PMID 33783365
- [Background] Small GW, Lee J, Kaufman A, Jalil J, Siddarth P, Gaddipati H, Moody TD, Bookheimer SY. Brain health consequences of digital technology use . Dialogues Clin Neurosci. 2020 Jun;22(2):179-187. doi: 10.31887/DCNS.2020.22.2/gsmall. PMID 32699518
- [Background] Scazufca M, Nakamura CA, Seward N, Didone TVN, Moretti FA, Oliveira da Costa M, Queiroz de Souza CH, Macias de Oliveira G, Souza Dos Santos M, Pereira LA, Mendes de Sa Martins M, van de Ven P, Hollingworth W, Peters TJ, Araya R. Self-help mobile messaging intervention for depression among older adults in resource-limited settings: a randomized controlled trial. Nat Med. 2024 Apr;30(4):1127-1133. doi: 10.1038/s41591-024-02864-4. Epub 2024 Mar 14. PMID 38486075
- [Background] Ngiam NHW, Yee WQ, Teo N, Yow KS, Soundararajan A, Lim JX, Lim HA, Tey A, Tang KWA, Tham CYX, Tan JPY, Lu SY, Yoon S, Ng KYY, Low LL. Building Digital Literacy in Older Adults of Low Socioeconomic Status in Singapore (Project Wire Up): Nonrandomized Controlled Trial. J Med Internet Res. 2022 Dec 2;24(12):e40341. doi: 10.2196/40341. PMID 36459398
- [Background] Mohamad Pilus F, Ahmad N, Mohd Zulkefli NA, Mohd Shukri NH. Effect of Face-to-Face and WhatsApp Communication of a Theory-Based Health Education Intervention on Breastfeeding Self-Efficacy (SeBF Intervention): Cluster Randomized Controlled Field Trial. JMIR Mhealth Uhealth. 2022 Sep 14;10(9):e31996. doi: 10.2196/31996. PMID 36103244
- [Background] Li Y, Shi H, Yuan Y, Zeng R, Bai B, Sun L. The impact of learning engagement on the subjective well-being of disadvantaged older adults in China. Front Public Health. 2023 Jul 18;11:1196692. doi: 10.3389/fpubh.2023.1196692. eCollection 2023. PMID 37533528
- [Background] Lee H, Lim JA, Nam HK. Effect of a Digital Literacy Program on Older Adults' Digital Social Behavior: A Quasi-Experimental Study. Int J Environ Res Public Health. 2022 Sep 29;19(19):12404. doi: 10.3390/ijerph191912404. PMID 36231707
- [Background] Chan MY, Haber S, Drew LM, Park DC. Training Older Adults to Use Tablet Computers: Does It Enhance Cognitive Function? Gerontologist. 2016 Jun;56(3):475-84. doi: 10.1093/geront/gnu057. Epub 2014 Jun 13. PMID 24928557
- [Background] Andre L, Giulioli C, Piau A, Bongard V, Richard E, Moll van Charante EP, Coley N, Andrieu S; PRODEMOS consortium. Telephone and Smartphone-Based Interventions for Cognitive and Cardio-Metabolic Health in Middle-Aged and Older Adults: A Systematic Review. Clin Interv Aging. 2022 Nov 10;17:1599-1624. doi: 10.2147/CIA.S352137. eCollection 2022. PMID 36393902
- See also: Older Singaporeans have low participation in learning. Programs show benefits but barriers remain, especially for socially disadvantaged groups. — https://www.duke-nus.edu.sg/docs/librariesprovider3/publications-docs/the-pursuit-of-learning-among-older-singaporeans.pdf?sfvrsn=24a70113_0